CLINICAL TRIAL: NCT05728450
Title: Effect of Laser Puncture on Liver Enzymes Post Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Lecturer of physical therapy of surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004203
Record Dates: First submitted 2023-01-19; First posted 2023-02-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: * The points for applying laser acupuncture will be cleaned before application. All patients in the study group will be submitted to an infrared diode laser, wavelength 808 nm, Pulse duration: 200 ms, Power density: 0.4 W/cm2, energy density 4 J/cm2 (Chow, 2001).
  * The plug of the laser unit will be inserted into the main current supply and the on/off switch will be switched on. The therapy form will be selected from the main menu and then the parameters will be set.
  * Acupuncture detector (Pointer Excel II) will be used for the actual location of acupuncture points.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): This group includes 15 burned patients who will receive laser puncture for one month (3 times/week) in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment.
  Interventions: Device: Light amplification by stimulated emission of radiation (LASER)
- Control group (No Intervention): This group includes 15 burned patients who will receive their physical therapy program (splinting, stretching ex., strengthening ex. and ROM ex.) and medical treatment.

INTERVENTIONS:
Device: Light amplification by stimulated emission of radiation (LASER) — * The points for application of laser acupuncture will be cleaned before application. All patients in the study group will be submitted to infrared diode laser, wavelength 808 nm, Pulse duration: 200 ms, Power density: 0.4 W/cm2, energy density 4 J/cm2 (Chow, 2001).
  * The plug of the laser unit will inserted into the main current supply and on/off switch will be switched on. The therapy form will be selected from the main menu and then the parameters will be set.
  * Acupuncture detector (Pointer Excel II) will be used for definite location of acupuncture points
  Arms: Study group

SUMMARY:
Procedures of laser puncture:

* The treatment procedures will start after the patient's release from the intensive care unit.
* The patient will be in a comfortable position.
* The patient will wear protective eyeglasses.
* The points for the application of laser acupuncture will be cleaned before application. All patients in the study group will be submitted to an infrared diode laser, wavelength 808 nm, Pulse duration: 200 ms, Power density: 0.4 W/cm2, energy density 4 J/cm2.
* The plug of the laser unit will be inserted into the main current supply and the on/off switch will be switched on. The therapy form will be selected from the main menu and then the parameters will be set.
* Acupuncture detector (Pointer Excel II) will be used for the definite location of acupuncture points.
* Laser probe will be placed in contact with the skin perpendicular over the body acupoints Zusanli (ST36), Taichong (LR3), Tanyinjiao (SP6), Ganshu (BL18), Yan-glingquan (GB34) and Zhongwan (RN12) in both sides, with a duration of 90 sec for each point three times per week for a month.

DETAILED DESCRIPTION:
Thirty patients with partial thickness burn with burned body surface area (BBSA) about 30% to 50% will participate in this study after their release from the intensive care unit. Their ages will be ranged from 20 to 45 years. The participants will be selected from Orabi hospital and randomly distributed into two equal groups.

1. Group A (Study group): This group includes 15 burned patients who will receive laser puncture for one month (3 times/week) in addition to their physical therapy program (splinting, stretching ex. and ROM ex.) and medical treatment.

1. Group B (Control group): This group includes 15 burned patients who will receive their physical therapy program (splinting, stretching ex., strengthening ex. and ROM ex.) and medical treatment.

Criteria for the patient selection:

- Inclusion Criteria:

The subject selection will be according to the following criteria:

* Age ranges between 20-45 years.
* Male and female patients will participate in the study.
* All patients who have burned with BBSA about 30% to 50% with acupoints are unaffected.
* All patients enrolled on the study will have their informed consent.
* Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Burn at areas of acupuncture points.
* Lower limb amputation.
* History of liver diseases.
* Body mass index (BMI=kg/cm2)<30%.

Procedures of laser puncture:

* The treatment procedures will start after the patient's release from the intensive care unit.
* The patient will be in a comfortable position.
* The patient will wear protective eyeglasses.
* The points for the application of laser acupuncture will be cleaned before application. All patients in the study group will be submitted to an infrared diode laser, wavelength 808 nm, Pulse duration: 200 ms, Power density: 0.4 W/cm2, energy density 4 J/cm2.
* The plug of the laser unit will be inserted into the main current supply and the on/off switch will be switched on. The therapy form will be selected from the main menu and then the parameters will be set.
* Acupuncture detector (Pointer Excel II) will be used for the definite location of acupuncture points.
* Laser probe will be placed in contact with the skin perpendicular over the body acupoints Zusanli (ST36), Taichong (LR3), Tanyinjiao (SP6), Ganshu (BL18), Yan-glingquan (GB34) and Zhongwan (RN12) in both sides, with a duration of 90 sec for each point three times per week for a month.

The anatomical locations of acupoints used:

1. Zusanli (ST36) acupoint is located on the lateral side of the lower leg, one hands' breadth below the knee crease and one finger's breadth lateral to the shin bone.
2. Tanyinjiao (SP6) acupoint is located on the inside of the lower leg, one hands' breadth above the prominence of the medial malleolus.
3. Taichong (LR3) acupoint is located on the dorsum of the foot in the distal hollow at the junction of the first and second metatarsal bone.
4. Yan-glingquan (GB34) acupoint is located below the outside of the knee, in a tender depression 1 body inch anterior and inferior to the head of the fibula.
5. Ganshu (BL18) acupoint is located two forefingers width lateral to the lower border of the spinous process of the 9th thoracic vertebra.
6. Zhongwan (RN12) acupoint is located on the anterior median line of the upper abdomen, proximal 5 fingers breadth above the belly button.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:
* Age ranges between 20-45 years.
* Male and female patients will participate in the study.
* All patients who have burned with BBSA about 30% to 50% with acupoints are unaffected.
* All patients enrolled on the study will have their informed consent.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* Burn at areas of acupuncture points.
* Lower limb amputation.
* History of liver diseases.
* Body mass index (BMI=kg/cm2)<30%.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-19 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
EFFECT OF LASER PUNCTURE ON LIVER ENZYMES POST BURN. | one month
  liver enzymes level (AST and ALT enzymes)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No